CLINICAL TRIAL: NCT04196777
Title: The Effect of Audit-and-feedback on the Excessive Use of Post-procedural Antimicrobials in Urologic Patients: a Pilot Intervention Study
Brief Title: Audit-and-feedback to Improve Antimicrobial-prescribing Among Urologists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Daniel Livorsi, Principal investigator, Iowa City Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 201911105
Record Dates: First submitted 2019-12-03; First posted 2019-12-12 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Urologic Diseases; Antibacterial Drug Adverse Reaction
Keywords: anti-bacterial
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Intervention Model Description: The behavioral intervention will be delivered at 3 intervention hospitals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): We will randomly select 3 intervention sites from the top quartile of all VHA sites, as ranked by the frequency of excessive post-procedural antimicrobial use after the 3 urologic procedures of interest. We will provide feedback both at baseline and at regular intervals to the 3 intervention sites. Data on hospital-level excessive post-procedural antimicrobial use specific to urologic patients (primary outcome) will be shared at baseline with the intervention sites. Updated data will be sent electronically to urology providers and the antimicrobial stewardship team at the intervention site every other month via electronic mail. These data will include an anonymous comparison to all other VHA hospitals.
  Interventions: Behavioral: Audit-and-feedback

INTERVENTIONS:
Behavioral: Audit-and-feedback — We will provide feedback both at baseline and at regular intervals to the 3 intervention sites. At first, we will schedule one-on-one conference calls with urology providers and the antimicrobial stewardship team at each of the 3 intervention sites. These conference calls will include a review of guidelines, a review of the facility's data on excessive post-procedural antimicrobial use for urologic patients, and an anonymous comparison to all other VHA sites. Next, we will prospectively monitor excessive post-procedural antimicrobial use at all 3 sites and the entire VHA for 1 year. Data on hospital-level excessive post-procedural antimicrobial use specific to urologic patients (primary outcome) will be sent electronically to urology providers and the antimicrobial stewardship team at the intervention site every other month via electronic mail.

SUMMARY:
Antimicrobial resistance is one of today''s most urgent public health problems. An important strategy to slow the spread of antimicrobial resistance is the promotion of judicious antimicrobial use. There are many opportunities to reduce unnecessary antimicrobial-prescribing, including in patients undergoing surgical procedures. The following study will specifically study opportunities to improve antimicrobial use in patients undergoing common urologic procedures at hospitals in the Veterans Health Administration (VHA).

Guidelines recommend giving antibiotics for no more than 24-hours after most urologic procedures, but the investigators have shown that the unnecessary use of post-procedural antimicrobials is common in this setting. In a national cohort of nearly 30,000 VHA patients, excessive post-procedural antimicrobials were prescribed after 37.2% of urologic procedures for a median duration of 3.0 excess days.

In this study, the investigators will evaluate whether giving regular feedback to providers at 3 VHA hospitals can reduce unnecessary antimicrobial use after urologic procedures.

DETAILED DESCRIPTION:
Trial design: The investigators propose a before/after quasi-experimental design, which will be analyzed with an interrupted time-series analysis.

Participants: There will be 3 intervention VHA hospitals. To be eligible, a VHA hospital must perform the following 3 urologic procedures: transurethral resection of the prostate (TURP), transurethral resection of a bladder tumor (TUBRT), and ureteroscopy (URS).

Interventions: The study team will conduct an audit-and-feedback intervention focused on the unnecessary use of prolonged antimicrobial therapy after common urologic procedures.

The audit-and-feedback intervention will target the urology providers at the 3 intervention sites.

Outcomes: The primary outcome for this study will be the frequency of excessive post-procedural antimicrobial-prescribing in the 3 urologic procedures of interest. Secondary outcomes include several safety outcomes, such as late antimicrobial prescriptions, return visits, mortality, C. difficile testing and C. difficile infection.

For each site, the pretest period will be the 2-years prior to the intervention. The intervention itself will last 1-year.

Selection of sites: Intervention sites will be randomly selected from the top quartile of all sites, as ranked on the frequency of excessive post-procedural antimicrobial-prescribing. If sites refuse to participate, additional sites will be invited until 3 sites agree to be enrolled.

Statistical methods: At the conclusion of the pilot trial, a quasi-experimental interrupted time-series (ITS) analysis will be performed to assess the change in monthly antimicrobial use for the 3 intervention sites combined. The time frame for this ITS analysis will be the two-years prior to the pilot trial's initiation through the trial's 1-year intervention period for a total of 36 months.

ELIGIBILITY:
Inclusion Criteria:

* A practicing urologist at an intervention site, OR
* A member of the antimicrobial stewardship team at an intervention site

Exclusion Criteria: None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - VA North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Iowa City VA Medical Center, Iowa City, Iowa
  - VA New York Harbor Healthcare System (Brooklyn), New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Livorsi DJ, Packiam VT, Shi Q, Alberding SY, Carter KD, Brown JA, Mason JB, Weiss JP, Steinberg RL. A pilot intervention trial to reduce the use of post-procedural antimicrobials after common endourologic surgeries. Infect Control Hosp Epidemiol. 2024 Nov 7;46(1):1-7. doi: 10.1017/ice.2024.172. Online ahead of print. PMID 39506499

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients who underwent a qualifying urologic procedure during 8/1/2022-7/31/2023 at a participating site were included in the intervention phase. These procedures were ureteroscopy (URS), transurethral resection of the prostate (TURP), and transurethral resection of a bladder tumor (TURBT). Outcomes in these enrolled patients were compared to outcomes in patients who underwent these qualifying procedures during a baseline period (n=1272); the baseline period spanned from 7/1/2020-6/30/2022.
Groups:
- Intervention: We will select 3 intervention sites that were above the median in their frequency of excessive post-procedural antimicrobial use after the 3 urologic procedures of interest, based on data from the 24-month baseline period. We will provide feedback both at baseline and at regular intervals to the 3 intervention sites. At first, we will schedule one-on-one conference calls with urology providers and the antimicrobial stewardship team at each of the 3 intervention sites. These conference calls will include a review of guidelines, a review of the facility's data on excessive post-procedural antimicrobial use for urologic patients, and an anonymous comparison to all other VHA sites. Next, we will prospectively monitor excessive post-procedural antimicrobial use at all 3 sites and the entire VHA for 1 year. Data on hospital-level excessive post-procedural antimicrobial use specific to urologic patients (primary outcome) will be sent electronically to urology providers and the antimicrobial stewardship team at the intervention site every other month via electronic mail. These data will include an anonymous comparison to all other VHA hospitals.
Period: Overall Study
Arm/Group | Intervention
Started | 525
Completed | 525
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline: Patients in the baseline group underwent one of the qualifying procedures at the 3 intervention sites during a period of time (7/1/2020-6/30/2022) before the intervention was implemented.
- Total: Total of all reporting groups
Arm/Group | Intervention | Baseline | Total
Number analyzed (Participants) | 525 | 1272 | 1797
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (10.4) | 71.6 (10.0) | 71.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 44 | 59
  Male | 510 | 1228 | 1738
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 36 | 55
  Not Hispanic or Latino | 455 | 1175 | 1630
  Unknown or Not Reported | 51 | 61 | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  Black or African American | 97 | 155 | 252
  White | 378 | 1026 | 1404
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 44 | 82 | 126
Transurethral resection of a bladder tumor [Count of Participants; unit: Participants] | 282 | 731 | 1013
Transurethral resection of prostate [Count of Participants; unit: Participants] | 130 | 260 | 390
Ureteroscopy [Count of Participants; unit: Participants] | 113 | 281 | 394

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cases Who Received Excessive Post-procedural Antimicrobials
Description: Excessive post-procedural antimicrobial use is defined as a prescription for a antimicrobial agent on post-procedural day one. For this specific outcome measure, the numerator will be the number of patients who received an excessive post-procedural antimicrobial, and the denominator will be all patients at the site who underwent a qualifying urologic procedure.
Time Frame: Within 1 day of the urologic procedure
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: This data shows the primary outcome during the 12-month audit-and-feedback period.
- Baseline Period: This data shows the primary outcome during the 24-month pre-intervention period.
Arm/Group | Intervention | Baseline Period
Number analyzed (Participants) | 525 | 1272
Participants | 216 | 644
Statistical Analysis 1: Comparison: Intervention vs Baseline Period; To model the primary outcome for site 3, we used a logistic regression model and a set of three explanatory variables: time, a binary indicator for an observation occurring within the intervention phase, and an interaction term between these two main effects (time and intervention); Test type: Other — We performed a logistic regression analysis that measured the effect of the intervention at site 3. The below results show the interaction term between time and the intervention from this model. Time was measured in days divided by 365, giving an annualized figure for the time coefficient estimate and interaction coefficient; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 0.089, 95% CI 2-sided [0.016 to 0.445]
Statistical Analysis 2: Comparison: Intervention vs Baseline Period; To model the primary outcome for site 1, we used a logistic regression model and a set of three explanatory variables: time, a binary indicator for an observation occurring within the intervention phase, and an interaction term between these two main effects (time and intervention); Test type: Other — We performed a logistic regression analysis that measured the effect of the intervention at site 1. The below results show the interaction term between time and the intervention from this model. Time was measured in days divided by 365, giving an annualized figure for the time coefficient estimate and interaction coefficient; p = 0.259, Regression, Logistic; Odds Ratio (OR) = 1.593, 95% CI 2-sided [0.710 to 3.585]
Statistical Analysis 3: Comparison: Intervention vs Baseline Period; To model the primary outcome for site 2, we used a logistic regression model and a set of three explanatory variables: time, a binary indicator for an observation occurring within the intervention phase, and an interaction term between these two main effects (time and intervention); Test type: Other — We performed a logistic regression analysis that measured the effect of the intervention at site 2. The below results show the interaction term between time and the intervention from this model. Time was measured in days divided by 365, giving an annualized figure for the time coefficient estimate and interaction coefficient; p = 0.738, Regression, Logistic; Odds Ratio (OR) = 0.748, 95% CI 2-sided [0.135 to 4.147]

2. Secondary Outcome: Excessive Post-procedural Antimicrobial Duration (Mean)
Description: Excessive post-procedural antimicrobial duration is defined as the duration of continuous excessive post-procedural antimicrobial use, as quantified as days of therapy per National Healthcare Safety Network methodology. This outcome will be calculated for each patient who underwent a qualifying procedure and received a post-procedural antimicrobial (primary outcome).
Time Frame: Within 30-days of the urologic procedure
Measure: Mean (Standard Deviation); unit: Days of antimicrobial therapy
Groups:
- Intervention: This data reflects the mean duration of excessive post-procedural antimicrobial use in patients who received post-procedural antimicrobials during the 12-month intervention period.
- Baseline: This data reflects the mean duration of excessive post-procedural antimicrobial use in patients who received post-procedural antimicrobials during the 24-month baseline period.
Arm/Group | Intervention | Baseline
Number analyzed (Participants) | 216 | 644
Days of antimicrobial therapy | 4.1 (6.4) | 5.3 (6.4)
Statistical Analysis 1: Comparison: Intervention; The median duration of post-procedural antimicrobial prescriptions at site 3 were compared using the Wilcoxon rank-sum test; Test type: Other — The Wilcoxon rank-sum test assessed whether the post-procedural antimicrobial duration significantly differed at site 3 between the baseline and intervention periods; p = 0.001, Wilcoxon (Mann-Whitney); Rank sum test statistic = 1280.5
Statistical Analysis 2: Comparison: Intervention vs Baseline; The median duration of post-procedural antimicrobial prescriptions at site 1 were compared using the Wilcoxon rank-sum test.Type of statistical test; Test type: Other — The Wilcoxon rank-sum test assessed whether the post-procedural antimicrobial duration significantly differed at site 1 between the baseline and intervention periods; p = 0.013, Wilcoxon (Mann-Whitney); Rank sum test statistic = 28662
Statistical Analysis 3: Comparison: Intervention vs Baseline; The median duration of post-procedural antimicrobial prescriptions at site 2 were compared using the Wilcoxon rank-sum test; Test type: Other — The Wilcoxon rank-sum test assessed whether the post-procedural antimicrobial duration significantly differed at site 2 between the baseline and intervention periods; p = 0.14, Wilcoxon (Mann-Whitney); Rank sum test statistic = 784

3. Secondary Outcome: Percentage of Cases Who Received a Late Antimicrobial Prescription
Description: Late antimicrobial prescription is defined as the prescription of a designated antimicrobial that does not qualify as a post-procedural antimicrobial (see above) by any provider within 7-30 days of the date of the patient's urologic procedure. For this specific outcome measure, the numerator will be the number of patients who received a late antimicrobial, and the denominator will be all patients at the site who underwent a qualifying urologic procedure.
Time Frame: Within 30-days of the urologic procedure
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: This data shows the proportion of cases who received a late antimicrobial prescription (see above definition) during the 12-month audit-and-feedback period.
- Baseline Period: This data shows the proportion of cases who received a late antimicrobial prescription (see above definition) during the 24-month pre-intervention period.
Arm/Group | Intervention | Baseline Period
Number analyzed (Participants) | 525 | 1272
Participants | 83 | 169
Statistical Analysis 1: Comparison: Intervention vs Baseline Period; To model this secondary outcome, we used a logistic regression model and a set of four explanatory variables: time, a binary indicator for an observation occurring within the intervention phase, an interaction term between these two main effects (time and intervention), and a binary indicator for the primary outcome. This last variable was included to assess the risk of these secondary outcomes in patients who were not exposed to post-procedural antimicrobials compared to those who were exposed; Test type: Other — We performed a logistic regression model that included patients across all 3 sites; p = 0.04, Regression, Logistic; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.58 to 0.99]

4. Secondary Outcome: Percentage of Cases Who Were Re-admitted to the Hospital or Presented to an Emergency Department or an Urgent Care Clinic
Description: Return visits: sought urgent/emergent healthcare for any indication within 30 days of the patient's index urologic procedure. For this specific outcome measure, the numerator will be the number of patients who had a return visit for any reason within 30-days of the urologic procedure, and the denominator will be all patients at the site who underwent a qualifying urologic procedure.
Time Frame: Within 30-days of the urologic procedure
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: This data shows the proportion of cases who had an unplanned visit (see above definition) during the 12-month audit-and-feedback period.
- Baseline Period: This data shows the proportion of cases who had an unplanned visit (see above definition) during the 24-month pre-intervention period.
Arm/Group | Intervention | Baseline Period
Number analyzed (Participants) | 525 | 1272
Participants | 113 | 186
Statistical Analysis 1: Comparison: Intervention vs Baseline Period; To model this secondary outcome across all sites, we used a logistic regression model and a set of four explanatory variables: time, a binary indicator for an observation occurring within the intervention phase, an interaction term between these two main effects (time and intervention), and a binary indicator for the primary outcome; Test type: Other — We performed a logistic regression model that included patients across all 3 sites; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.53 to 0.87]

5. Secondary Outcome: Percentage of Cases Who Died (Mortality)
Description: Mortality: all-cause death within 30-days of the patient's index urologic procedure. For this specific outcome measure, the numerator will be the number of patients who died for any reason within 30-days of the urologic procedure, and the denominator will be all patients at the site who underwent a qualifying urologic procedure.
Time Frame: Within 30-days of the urologic procedure
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: This data shows the proportion of patients who died within 30 days after the procedure during the 12-month audit-and-feedback period.
- Baseline Period: This data shows the proportion of patients who died within 30 days after the procedure during the 24-month pre-intervention period.
Arm/Group | Intervention | Baseline Period
Number analyzed (Participants) | 525 | 1272
Participants | 4 | 4

6. Secondary Outcome: Percentage of Cases Who Underwent Clostridioides Difficile Testing
Description: Clostridioides difficile testing is defined as any laboratory test ordered for C. difficile within 30-days of the patient's urologic procedure. For this specific outcome measure, the numerator will be the number of patients who underwent C. difficile testing within 30-days of the procedure, and the denominator will be all patients at the site who underwent a qualifying urologic procedure.
Time Frame: Within 30-days of the urologic procedure
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: This data shows the proportion of cases who had C. difficile testing within 30 days after the procedure during the 12-month audit-and-feedback period.
- Baseline Period: This data shows the proportion of cases who had C. difficile testing within 30 days after the procedure during the 24-month pre-intervention period.
Arm/Group | Intervention | Baseline Period
Number analyzed (Participants) | 525 | 1272
Participants | 1 | 6

7. Secondary Outcome: Percentage of Cases Who Acquired Clostridioides Difficile Infection
Description: Clostridioides difficile infection (CDI) is defined as a positive laboratory test for C.difficile within 30-days of the patient's urologic procedure. For this specific outcome measure, the numerator will be the number of patients who had a positive test for C. difficile within 30-days of the procedure, and the denominator will be all patients at the site who underwent a qualifying urologic procedure.
Time Frame: Within 30-days of the urologic procedure
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: This data shows the proportion of cases who had a positive C. difficile test result within 30 days after the procedure during the 12-month audit-and-feedback period.
- Baseline Period: This data shows the proportion of cases who had a positive C. difficile test result within 30 days after the procedure during the 24-month pre-intervention period.
Arm/Group | Intervention | Baseline Period
Number analyzed (Participants) | 525 | 1272
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: We monitored for adverse events during the 30-day period after the qualifying procedure was performed.
Groups:
- Intervention: We will select 3 intervention sites who are above the median in their frequency of excessive post-procedural antimicrobial use after the 3 urologic procedures of interest, based on each hospital's performance during a 24-month baseline period. We will provide feedback both at baseline and at regular intervals to the 3 intervention sites. At first, we will schedule one-on-one conference calls with urology providers and the antimicrobial stewardship team at each of the 3 intervention sites. These conference calls will include a review of guidelines, a review of the facility's data on excessive post-procedural antimicrobial use for urologic patients, and an anonymous comparison to all other VHA sites. Next, we will prospectively monitor excessive post-procedural antimicrobial use at all 3 sites and the entire VHA for 1 year. Data on hospital-level excessive post-procedural antimicrobial use specific to urologic patients (primary outcome) will be sent electronically to urology providers and the antimicrobial stewardship team at the intervention site every other month via electronic mail. These data will include an anonymous comparison to all other VHA hospitals.
- Baseline: Adverse events were measured among patients who underwent a qualifying procedure at the 3 intervention sites prior to implementation of the intervention. This period spanned from 7/1/2020-6/30/2022.
Arm/Group | Intervention | Baseline
All-Cause Mortality (participants affected / at risk) | 4/525 | 4/1272
Serious Adverse Events (participants affected / at risk) | 113/525 | 186/1272
Other Adverse Events (participants affected / at risk) | 0/525 | 0/1272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=525) | Baseline (N=1272)
Emergency Department, Urgent Care Clinic, or Hospital Re-admission within 30 days of the procedure (Surgical and medical procedures) | 113 (113) | 186 (186) — The patient sought care in an Emergency Department, Urgent Care Clinic or hospital readmission to an acute-care bed at a VHA facility for any indication within 30 days of the patient's index urologic procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT04196777/Prot_SAP_000.pdf